CLINICAL TRIAL: NCT06708377
Title: Comparison of Effects Of Dry Needling And Myofascial Massage Therapy On Masseter Muscle In Patients With Temporomandibular Joint Dysfunction
Brief Title: Dry Needling and Myofascial Massage Therapy on Patient With Temporomandibular Joint Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Samiullah Khan
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Temporomandibular Joint Dysfunction
Keywords: TMJ Dysfunction; Dry needling; Myofascial massage therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling of masseter muscle (Experimental): Experimental group included Dry needling of masseter muscle for 30 second to 2 minutes into the trigger point.
  Conventional heating pad or face pad for 15 minutes. Therapeutic ultrasound with Frequency: 3MHz, Intensity: 0.75 - 1 W/cm2, Time: Based on treatment head and pulse factor. Temporomandibular joint mobilization (Maitland)-caudal glide, anterior-posterior glide, grade II, III, IV 3 reps x 3 sets per session. 6 x 6 exercise protocol of Rocabado, 6 reps per exercise x 6/day.
  Interventions: Other: dry needling of masseter
- Myofacial massage therapy (Active Comparator): Control group included Myofascial massage - sliding and kneading, for 30 minutes per session/3x per week. Conventional heating pad or face pad for 15 minutes. Therapeutic ultrasound with Frequency: 3MHz, Intensity: 0.75 - 1 W/cm2, Time: Based on treatment head and pulse factor. Temporomandibular joint mobilization (Maitland)-caudal glide, anterior-posterior glide, grade II, III, IV 3 reps x 3 sets per session. 6 x 6 exercise protocol of Rocabado, 6 reps per exercise x 6/day.
  Interventions: Other: myofascial massage therapy on masseter muscle

INTERVENTIONS:
Other: dry needling of masseter — Experimental group included Dry needling of masseter muscle for 30 second to 2 minutes into the trigger point.
  Conventional heating pad or face pad for 15 minutes. Therapeutic ultrasound with Frequency: 3MHz, Intensity: 0.75 - 1 W/cm2, Time: Based on treatment head and pulse factor. Temporomandibular joint mobilization (Maitland)-caudal glide, anterior-posterior glide, grade II, III, IV 3 reps x 3 sets per session. 6 x 6 exercise protocol of Rocabado, 6 reps per exercise x 6/day.
  Arms: Dry needling of masseter muscle
Other: myofascial massage therapy on masseter muscle — Control group included Myofascial massage - sliding and kneading, for 30 minutes per session/3x per week. Conventional heating pad or face pad for 15 minutes. Therapeutic ultrasound with Frequency: 3MHz, Intensity: 0.75 - 1 W/cm2, Time: Based on treatment head and pulse factor. Temporomandibular joint mobilization (Maitland)-caudal glide, anterior-posterior glide, grade II, III, IV 3 reps x 3 sets per session. 6 x 6 exercise protocol of Rocabado, 6 reps per exercise x 6/day
  Arms: Myofacial massage therapy

SUMMARY:
Comparison of effects of dry needling and myofascial massage therapy on masseter muscle in patients with temporomandibular joint dysfunction. A randomized control trial was conducted at DSK Physio & Rehab Centre, Ulfat Dental Associates and The Physiotherapy Clinic, Islamabad. The sample size was 24 calculated through G-power 3.1. The participants were divided into two interventional groups each having 12 participants. The study duration was six months. Sampling technique applied was convenience sampling for recruitment and group randomization using flip coin method. Only 25 to 45 years participants with having TMJ Dysfunction and reduced mouth opening were included in the study. Tools used in this study are NPRS, Maximal Mouth Opening and Fonseca Anamnestic Index. Data was collected at baseline, at the end of 1st week and 3rd week. Data analyzed through SPSS version26.

DETAILED DESCRIPTION:
Temporomandibular joint (TMJ) dysfunction encompasses a range of conditions affecting the jaw joint and surrounding muscles, often resulting in pain, restricted movement, and functional impairment. Temporomandibular disorder (TMD) can be categorized as intra-articular, affecting structures within the temporomandibular joint (TMJ), or extra-articular, involving surrounding muscles and structures. Intra-articular TMD includes conditions like disc displacement, osteoarthritis, or subluxation, while extra-articular TMD manifests as muscle pain or dysfunction, such as myofascial pain syndrome.

Reduced mouth opening or limited mandibular range of motion, is a condition characterized by restricted movement of the TMJ resulting in diminished ability to open the mouth. It can arise from various etiologies including trauma, inflammation, muscle dysfunction, or surgical interventions affecting the masticatory muscles or TMJ. Trismus may manifest acutely or chronically and can significantly impair oral functions such as eating, speaking, and oral hygiene maintenance. Assessment typically involves measurement of maximal inter-incisal opening (MIO) using standardized methods, with normal values varying depending on age, gender, and population.

The Maximal Mouth Opening (MMO) generalized reference range is from 42 to 60 mm.

Patients diagnosed with myofascial temporomandibular disorder (TMD) commonly present myofascial trigger points (MTrPs) located in both the neck and masticatory muscles. These trigger points are believed to be integral to the development and expression of myofascial TMD symptoms. MTrPs represent hypersensitive sites within taut bands of skeletal muscle or muscle fascia. Their activation can lead to a range of sensory, motor, neurological, and autonomic symptoms, contributing significantly to the clinical presentation of myofascial TMD. Among the various treatment modalities, myofascial massage therapy and dry needling have gained attention for their potential efficacy in managing TMJ dysfunction, particularly in addressing the associated muscular component.

Myofascial massage therapy targets the fascia, the connective tissue surrounding muscles, aiming to release tension, improve blood flow, and restore mobility. Massage therapy can help break down trigger points through several mechanisms. Firstly, it increases blood flow to the affected area, which helps deliver oxygen and nutrients while removing waste products, aiding in tissue repair. It can also disrupt the tight muscle fibers and release tension, allowing the muscle to relax and the trigger point to dissipate. Additionally, massage stimulates the nervous system, promoting the release of endorphins and other natural pain-relieving chemicals, which can help alleviate discomfort associated with trigger points. Lastly, the pressure and manipulation applied during massage can physically break down adhesions and knots within the muscle tissue, helping to release the trigger point.In the context of TMJ dysfunction, myofascial massage may involve techniques such as effleurage, petrissage, and trigger point therapy to alleviate muscle tightness, reduce pain, and enhance jaw function.

This approach focuses on manual manipulation of soft tissues to promote relaxation and alleviate muscular imbalances contributing to TMJ symptoms. Dry needling involves the insertion of thin needles into trigger points or areas of muscular tension to elicit a therapeutic response. Unlike acupuncture, which follows traditional Chinese medicine principles, dry needling targets specific muscular trigger points rather than meridian pathways.

In the context of TMJ dysfunction, dry needling aims to deactivate hyperirritable trigger points, reduce muscle tension, and alleviate pain by promoting local blood flow and releasing endogenous opioids. The recent systematic review emphasized the necessity for conducting larger trials with a decreased risk of bias to thoroughly evaluate the impact of dry needling on myofascial temporomandibular disorder (TMD). This recommendation stems from the observation of both the low quality of evidence and the heightened risk of bias evident in certain studies included in the review.

While both myofascial massage therapy and dry needling target muscular dysfunction associated with TMJ disorders, they differ in their mechanisms of action and application. Myofascial massage therapy relies on manual manipulation techniques to directly address muscle tension and fascial restrictions, promoting relaxation and improved tissue mobility. In contrast, dry needling involves the precise insertion of needles into trigger points to stimulate neuromuscular responses and induce therapeutic effects, such as pain relief and muscle relaxation. Dry needling is a common intervention in clinical practice nowadays, but its effectiveness compared to other conservative treatment modalities, such as manual therapy, remains unclear.

In a 2022 network meta-analysis (NMA), which evaluated the effectiveness of twelve different treatment modalities for patients with myofascial temporomandibular disorder (TMD), manual therapy emerged as the most effective treatment option. Nevertheless, the authors advised a careful interpretation of the findings, citing study limitations and a paucity of robust evidence.

According to a systematic review published in 2023, it was concluded that no significant differences in terms of pain reduction was observed between dry needling and manual therapy in patients with myofascial TMD. High variability was observed in available literature for methods of application of these interventions.

Despite growing interest in myofascial massage therapy and dry needling for TMJ dysfunction, there remains a gap in the literature regarding direct comparisons of their efficacy, safety, and long-term outcomes. While individual studies have investigated the effects of each modality separately, few studies have directly compared their effectiveness in improving TMJ symptoms and functional outcomes. Additionally, factors such as treatment protocols, patient characteristics, and practitioner expertise may influence treatment outcomes and complicate direct comparisons between myofascial massage therapy and dry needling.

This lack of comparative randomized clinical trials between dry needling and myofascial massage therapy limits determine which technique of the two is better. So, the available literature has only made indirect comparisons and therefore, the current study aims to find the comparative effectiveness of myofascial massage therapy and dry needling for TMJ dysfunction. The findings will help inform evidence-based management strategies for TMJ dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Participants with TMJ dysfunction
* A mouth opening of less than 39 mm for males and 36mm for females
* Patients with Trigger points in tout band of masseter
* Mild to moderate pain on NPRS
* 45-75 points on Fonseca's questionnaire

Exclusion Criteria:

* Bell's palsy
* Trigeminal neuralgia
* Wearing any form of dental prosthesis
* Any form of surgery in or around the TMJ
* History of trauma or fracture in and around the TMJ
* Not consenting to take part in the study

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-12-03 (Estimated); Study Completion 2024-12-13 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 5 mints at every session
  changes from the baseline pain intensity was measured using numeric pain rating scale
Maximum Mouth Opening (MMO) | 10 mint at every session
  changes from baseline maximum mouth opening were measured in mm using fiber ruler

SECONDARY OUTCOMES:
Fonseca Anamnestic Index (FAI) | 15 mints
  changes from baseline TMJ Dysfunction was measured using FAI

CONTACTS AND LOCATIONS:
Overall Officials: Lal Gul Khan, MScPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poveda Roda R, Diaz Fernandez JM, Hernandez Bazan S, Jimenez Soriano Y, Margaix M, Sarrion G. A review of temporomandibular joint disease (TMJD). Part II: Clinical and radiological semiology. Morbidity processes. Med Oral Patol Oral Cir Bucal. 2008 Feb 1;13(2):E102-9. PMID 18223525
- [Background] Okeson JP. Joint intracapsular disorders: diagnostic and nonsurgical management considerations. Dent Clin North Am. 2007 Jan;51(1):85-103, vi. doi: 10.1016/j.cden.2006.09.009. PMID 17185061
- [Background] Chaudhary F, Ahmad B, Butt D, Hameed S, Bashir U. Normal range of maximum mouth opening in pakistani population: A cross-sectional study. Journal of International Oral Health. 2019;11:353
- [Background] Fernandez-de-Las-Penas C, Galan-Del-Rio F, Alonso-Blanco C, Jimenez-Garcia R, Arendt-Nielsen L, Svensson P. Referred pain from muscle trigger points in the masticatory and neck-shoulder musculature in women with temporomandibular disoders. J Pain. 2010 Dec;11(12):1295-304. doi: 10.1016/j.jpain.2010.03.005. Epub 2010 May 21. PMID 20494623
- [Background] Travell JG SD. Myofascial pain and dysfunction: the trigger point manual. Lippincott Williams & Wilkins. 1992.
- [Background] Medlicott MS, Harris SR. A systematic review of the effectiveness of exercise, manual therapy, electrotherapy, relaxation training, and biofeedback in the management of temporomandibular disorder. Phys Ther. 2006 Jul;86(7):955-73. PMID 16813476
- [Background] Vier C, Almeida MB, Neves ML, Santos ARSD, Bracht MA. The effectiveness of dry needling for patients with orofacial pain associated with temporomandibular dysfunction: a systematic review and meta-analysis. Braz J Phys Ther. 2019 Jan-Feb;23(1):3-11. doi: 10.1016/j.bjpt.2018.08.008. Epub 2018 Aug 22. PMID 30146108
- [Background] Leeuw R. Orofacial pain: Guidelines for assessment, diagnosis, and management. Chicago: American Academy of Orofacial. 2008:1-24.
- [Background] Menendez-Torre A, Pintado-Zugasti AM, Zaldivar JNC, Garcia-Bermejo P, Gomez-Costa D, Molina-Alvarez M, Arribas-Romano A, Fernandez-Carnero J. Effectiveness of deep dry needling versus manual therapy in the treatment of myofascial temporomandibular disorders: a systematic review and network meta-analysis. Chiropr Man Therap. 2023 Nov 3;31(1):46. doi: 10.1186/s12998-023-00489-x. PMID 37924127
- [Background] Al-Moraissi EA, Conti PCR, Alyahya A, Alkebsi K, Elsharkawy A, Christidis N. The hierarchy of different treatments for myogenous temporomandibular disorders: a systematic review and network meta-analysis of randomized clinical trials. Oral Maxillofac Surg. 2022 Dec;26(4):519-533. doi: 10.1007/s10006-021-01009-y. Epub 2021 Oct 21. PMID 34674093
- [Background] Dib-Zakkour J, Flores-Fraile J, Montero-Martin J, Dib-Zakkour S, Dib-Zaitun I. Evaluation of the Effectiveness of Dry Needling in the Treatment of Myogenous Temporomandibular Joint Disorders. Medicina (Kaunas). 2022 Feb 9;58(2):256. doi: 10.3390/medicina58020256. PMID 35208580
- [Background] Chiarotto A, Maxwell LJ, Ostelo RW, Boers M, Tugwell P, Terwee CB. Measurement Properties of Visual Analogue Scale, Numeric Rating Scale, and Pain Severity Subscale of the Brief Pain Inventory in Patients With Low Back Pain: A Systematic Review. J Pain. 2019 Mar;20(3):245-263. doi: 10.1016/j.jpain.2018.07.009. Epub 2018 Aug 10. PMID 30099210
- [Background] Nomura K, Vitti M, Oliveira AS, Chaves TC, Semprini M, Siessere S, Hallak JE, Regalo SC. Use of the Fonseca's questionnaire to assess the prevalence and severity of temporomandibular disorders in Brazilian dental undergraduates. Braz Dent J. 2007;18(2):163-7. doi: 10.1590/s0103-64402007000200015. PMID 17982559
- [Background] Zagalaz-Anula N, Sanchez-Torrelo CM, Acebal-Blanco F, Alonso-Royo R, Ibanez-Vera AJ, Obrero-Gaitan E, Rodriguez-Almagro D, Lomas-Vega R. The Short Form of the Fonseca Anamnestic Index for the Screening of Temporomandibular Disorders: Validity and Reliability in a Spanish-Speaking Population. J Clin Med. 2021 Dec 14;10(24):5858. doi: 10.3390/jcm10245858. PMID 34945153
- [Background] Gerwin RD, Shannon S, Hong CZ, Hubbard D, Gevirtz R. Interrater reliability in myofascial trigger point examination. Pain. 1997 Jan;69(1-2):65-73. doi: 10.1016/s0304-3959(96)03248-4. PMID 9060014
- [Background] Lew J, Kim J, Nair P. Comparison of dry needling and trigger point manual therapy in patients with neck and upper back myofascial pain syndrome: a systematic review and meta-analysis. J Man Manip Ther. 2021 Jun;29(3):136-146. doi: 10.1080/10669817.2020.1822618. Epub 2020 Sep 22. PMID 32962567
- [Background] Biasotto-gonzalez DA. Abordagem interdisciplinar das disfunções temporomandibulares: Editora Manole Ltda; 2005.
- [Background] Gomes CA, Politti F, Andrade DV, de Sousa DF, Herpich CM, Dibai-Filho AV, Gonzalez Tde O, Biasotto-Gonzalez DA. Effects of massage therapy and occlusal splint therapy on mandibular range of motion in individuals with temporomandibular disorder: a randomized clinical trial. J Manipulative Physiol Ther. 2014 Mar-Apr;37(3):164-9. doi: 10.1016/j.jmpt.2013.12.007. Epub 2014 Jan 3. PMID 24387891